CLINICAL TRIAL: NCT04280458
Title: Impact of Intensive Psychomotor Rehabilitation on Cognitive-motor Abilities and Adaptive Capacity of Children With Polyhandicap
Brief Title: Intensive Psychomotor Rehabilitation on Cognitive Motor Abilities and Adaptive Capacity on Children With Polyhandicap
Acronym: REEDUC-PLH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: APHP200866; 2020-A00800-39 (Registry Identifier: IDRCB)
Record Dates: First submitted 2020-02-17; First posted 2020-02-21 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Polyhandicap
Keywords: children polyhandicap; rehabilitation; psychomotor; cognitive-motor; adaptative skill

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): patients will receive intensive care of rehabilitation of psychomotor
  Interventions: Behavioral: Intentive rehabilitation
- Control group (Active Comparator): patients will receive standard care
  Interventions: Behavioral: Routine care

INTERVENTIONS:
Behavioral: Intentive rehabilitation — Intervention included:
  * psychomotor 5 hours/week ±30 minutes
  * kinesitherapy 1.5 hour/week ±20 minutes
  during 12 months.
  Arms: Intervention group
Behavioral: Routine care — Intervention included:
  * kinesitherapy 0.5 hour/week ±10 minutes
  * psychomotor 30 min/week ±10 minutes during 12 months.
  Arms: Control group

SUMMARY:
Primary objective of the study is to compare and evaluate the impact of intensive care of rehabilitation of psychomotor vs. the standard care on adaptive behaviour of children with polyhandicap at 12 months after randomization.

DETAILED DESCRIPTION:
As secondary objectives, the study aims to:

1. compare and evaluate the impact of this intensive care of rehabilitation of psychomotor vs. the standard care on:

   * result of evaluation with Vineland Scale of adaptive behaviour at 6 months after randomization;
   * result of evaluation with Brunet-Lézine Scale of developement at 12 months after randomization;
   * the pain evaluation at 12 months after randomization;
   * the durability of acquired cognitive-motor improvement at 6 months after the end of intervention (18 months after randomization);
   * the quality of life of the patients' family or relatives at 12 months after randomization;
   * the clinical global impressions and the quality of life for work for the long-term professional caregivers at 12 months after randomization.
2. evaluate the tolerance of intensive care in psychomotor rehabilitation at 6 and 12 months after randomization.
3. study the concordance between the Vineland scale and the Brunet-Lézine scale.

ELIGIBILITY:
Inclusion Criteria:

* Children between 4 and 13 years;
* With polyhandicap defined by association of the 5 following criteria:

  * Causal brain injury occurred before the age of 3 years
  * Severe or deep mental deficiency as defined by IQ < 40, or no evaluable by the psychometric tests
  * Motor impairment: para / tetraparesis, hemiparesis, ataxia, or extrapyramidal motor disorders
  * Score of Gross Motor Function Classification System [Palisano 1997] is III, IV or V
  * Score of Functional Independence Measure < 50;
* Hospitalization in a clinical setting participating to the study;
* Beneficiary of a social protection;
* Written consent signed by personnel holding parental authority or legal representative.

Exclusion Criteria:

* Patient with progressive encephalopathies including metabolic origin, epileptic, or neurodegenerative diseases;
* Planned to move in another clinical setting;
* Foreseeable difficulty in the following up in the study.

Ages: 4 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Estimated)
Dates: Start 2022-06-20 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of adaptative behaviour | At 12 months
  Vineland II Scale will be used to evaluate the evolution of adaptative behaviour.

SECONDARY OUTCOMES:
Evolution of adaptative behaviour | At 6 months
  Vineland II Scale will be used to evaluate the evolution of adaptative behaviour.
Evolution of development | At 12 months
  Brunet-Lézine Scale will be used to evaluate the evolution of development.
Pain evaluation | At 12 months
  Scale named Echelle Douleur Enfant San Salvadour (EDESS, in French language) will be used to evaluate the pain.
Durability of acquired cognitive-motor abilities | at 18 months
  Vineland Adaptativ Behavior Scales will be used to evaluate durability of acquired cognitive-motor abilities.
Durability of acquired cognitive-motor abilities | at 18 months
  The Brunet-Lézine scale for the cognitive and motor assessment will be used to evaluate durability of acquired cognitive-motor abilities.
Quality of family's life surveys | At baseline and 12 months
  WHOQOL-Bref questionnaire will be used.
Emotional distress measurement | At baseline and 12 months
  Hospital Anxiety and Depression Scale will be used to evaluate the emotional distress of polyhandicapped children's parents.
Burden surveys | At baseline and 12 months
  Caregiver Reaction Assessment (CRA) will be used to evaluate the specific burden of polyhandicapped children's parents.
Clinical Global Impressions by caregivers | At baseline and 12 months
  Clinical Global Impressions (CGI) Scale will be used by caregivers.
Quality of caregivers' life | At baseline and 12 months
  The tool as Professional Quality of Life ProQOL will be used to measure quality of life of caregivers.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Christine ROUSSEAU, MD, Principal Investigator — Polyhandicap adultes San Salvadour, APHP
Locations (1):
- Hôpital San Salvadour, Hyères, Var, France

REFERENCES:
- [Background] Collignon P, Giusiano B. Validation of a pain evaluation scale for patients with severe cerebral palsy. Eur J Pain. 2001;5(4):433-42. doi: 10.1053/eujp.2001.0265. PMID 11743709
- [Background] Busner J, Targum SD. The clinical global impressions scale: applying a research tool in clinical practice. Psychiatry (Edgmont). 2007 Jul;4(7):28-37. PMID 20526405
- [Background] Laor-Maayany R, Goldzweig G, Hasson-Ohayon I, Bar-Sela G, Engler-Gross A, Braun M. Compassion fatigue among oncologists: the role of grief, sense of failure, and exposure to suffering and death. Support Care Cancer. 2020 Apr;28(4):2025-2031. doi: 10.1007/s00520-019-05009-3. Epub 2019 Aug 8. PMID 31392551